CLINICAL TRIAL: NCT02414997
Title: The Effect of Remote Ischemic Preconditioning (RIPC) on Blood Pressure and Its Vascular Protection Effect Among Chinese Young Healthy Adults and Primary Hypertensive Patients Stage I
Brief Title: The Effect of Remote Ischemic Preconditioning (RIPC) on Blood Pressure and Its Vascular Protection Effect
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiao Haipeng, president, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHaipeng
Record Dates: First submitted 2015-03-27; First posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Pressure; Brachial Plexus
Keywords: RIPC (remote ischemic preconditioning); primary hypertension stage I; vascular function; microRNA-126; microRNA-34a
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC group (Experimental): Surround left upper limb with cuff, inflate cuff to 200 mmHg and maintain 5 minutes, than deflate to 0 mmHg. Change to right upper limb and repeat the procedure described above. Change back to left upper limb and repeat the same procedure. Perform once a day ( Thus 15 minutes a day).
  Interventions: Procedure: RIPC
- Sham RIPC group (Sham Comparator): Surround left upper limb with cuff, inflate cuff to 20 mmHg and maintain 5 minutes, than deflate to 0 mmHg. Change to right upper limb and repeat the procedure described above. Change back to left upper limb and repeat the same procedure. Perform once a day ( Thus 15 minutes a day).
  Interventions: Procedure: Sham RIPC

INTERVENTIONS:
Procedure: RIPC — Surround left upper limb with cuff, inflate cuff to 200mmHg and maintain 5 minutes, than deflate to 0mmHg. Change to right upper limb and repeat the procedure described above. Change back to left upper limb and repeat the same procedure. Perform once a day ( Thus 15 minutes a day).
  Arms: RIPC group
Procedure: Sham RIPC — Surround left upper limb with cuff, inflate cuff to 20mmHg and maintain 5 minutes, than deflate to 0mmHg. Change to right upper limb and repeat the procedure described above. Change back to left upper limb and repeat the same procedure. Perform once a day ( Thus 15 minutes a day).
  Arms: Sham RIPC group

SUMMARY:
The purpose of this study is to determine the effect of remote ischemic preconditioning (RIPC) on blood pressure and its vascular protection effect among Chinese young healthy adults and primary hypertensive patients stage I.

DETAILED DESCRIPTION:
Hypertension is one of the most common world-wide chronic diseases, and it is one of major independent risk factors of atherosclerotic cardiovascular diseases (ASCVD) especially among middle-aged and elderly. Recently, a study indicates that in a normotensive elderly without cardiovascular diseases history, continuous RIPC for 30 days lowers systolic blood pressure for 6 mmHg and diastolic blood pressure for 3 mmHg. Another study shows a 7-day RIPC intervention improves endothelium-dependent flow mediated dilation(FDM) and cutaneous vascular conductivity(CVC) in 13 healthy young males. In addition, studies demonstrate that microRNA-126 and microRNA-34a are endothelial specific microRNAs which are expressed in human PBMCs. MicroRNA-126 is responsible for keeping the integrity of vascular endothelial, promoting the proliferation, mobilization, and migration of endothelial progenitor cells(EPCs), reducing arterial intimal hyperplasia, and reduce adhesion of neutrophils to vascular endothelial. In contrast, microRNA-34a is related to the aging of endothelial cells, which is found over-expressed in senile endothelial cells. Together the investigators use microRNA-126 and microRNA-34a to explore whether RIPC produces vascular endothelial protection effect. In summary, the investigators propose a hypothesis that RIPC might have a blood pressure lowing effect and protect vascular function both in Chinese healthy young adults and primary hypertensive patients. The term "primary hypertension stage I" indicates those with blood pressures ranging from 140 to 159 mmHg systolic and/or 90 to 99 mmHg diastolic. Accumulating evidences suggest that subjects with primary hypertension stage I are associated with higher incidence of ASCVD. However, there is no available data to investigate a nonpharmacologic therapy for primary hypertension stage I until now, and there is no prospective, randomized, controlled, single-blind clinic trial to investigate the effect of RIPC on blood pressure and its vascular protection effect. The investigators hypothesize that RIPC may lower both SBP and DBP, and it improves vascular function in Chinese healthy young adults and subjects with primary hypertension stage I. To address these assumptions, the present study is designed to study the effect of RIPC on blood pressure and its vascular protection effect, using FMD, PWV, central arterial pressure, RHI(EndoPAT) and the quantification of microRNA-126 and microRNA-34a in peripheral blood monocyte(PBMC) as indicators among Chinese healthy young adults and primary hypertensive patients stage I over a 1-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects range from 18 to 80 years old.
* Blood pressure is normal or primary hypertension stage I(systolic blood pressure 140 to 159 mmHg and/or diastolic blood pressure 90 to 99 mmHg).
* No history of smoking( smoking can eliminate the effect of RIPC) or quit smoking for at least 1 years.
* No intake of caffeine or caffeine-containing substances during the process of this trial(caffeine can eliminate the effect of RIPC).
* Provide informed consent and willingness to cooperate with the study protocol.

Exclusion Criteria:

* Less than 18 years old or above 80 years old.
* Secondary hypertension.
* Pregnant or lactating females.
* Systemic diseases such as diabetes, HIV/AIDS, liver disease, chronic renal failure, tuberculosis, and autoimmune diseases.
* Medical history of cardiovascular disease: acute myocardial infarct, stable angina, unstable angina, heart failure, atrial fibrillation, atrioventricular blockade, peripheral vascular disease or cerebrovascular accident.
* Patients who are unfavorable of long-term follow-up or poor compliance.
* Patients who are considered unfavorable to take part in this trial by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure at 1 month | Baseline; 1 week after RIPC; 1 month after RIPC
  systolic pressure lowers 6mmHg
Change from Baseline in Diastolic Blood Pressure at 1 month | Baseline; 1 week after RIPC; 1 month after RIPC
  diastolic pressure lowers 3mmHg

SECONDARY OUTCOMES:
Artery elasticity | Baseline; 1 week after RIPC; 1 month after RIPC
  Brachia-ankle pulse wave velocity (baPWV)
Vascular endothelial function - RHI(EndoPAT) | Baseline; 1 week after RIPC; 1 month after RIPC
  RHI
Quantification of microRNA-126 and microRNA-34a in PBMC (peripheral blood mononuclear cell) | Baseline; 1 week after RIPC; 1 month after RIPC
Migration and adhesion function of endothelial progenitor cells (EPC) | Baseline; 1 week after RIPC; 1 month after RIPC
Endothelial function | Baseline; 1 week after RIPC; 1 month after RIPC
  Endothelium-dependent brachial artery flow-mediated dilation (FMD)
Expression of CXC-chemokine receptor 4 and CXC-chemokine receptor 7 protein of EPC | Baseline; 1 week after RIPC; 1 month after RIPC

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jun, phD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University